CLINICAL TRIAL: NCT02151864
Title: Phase Ib Study of Single Agent LDE225, an Oral Hedgehog Inhibitor, as Second-Line Therapy in Patients With Advanced or Metastatic Hepatocellular Carcinoma and Child-Pugh A/B7 Cirrhosis
Brief Title: LDE225 in Patients With Advanced or Metastatic Hepatocellular Carcinoma and Child-Pugh A/B7 Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jason K. Sicklick, M.D. (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jason K. Sicklick, M.D., Assistant Professor, Surgery, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 131053
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: liver cancer; cirrhosis; Child-Pugh A; Hedgehog
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Liver Neoplasms | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LDE225 (Experimental): LDE225 200mg-800mg oral daily
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — LDE225 will be administered orally, on a continuous once daily dosing schedule at a dose determined by the cohort the patient is enrolled in until progression or unacceptable toxicity develops
  Other Names: hedgehog inhibitor

SUMMARY:
The purpose of this study is to test the safety and determine the maximum safe dose of an experimental drug called LDE225 (hedgehog inhibitor) in people with liver cancer. We have identified hedgehog dysregulation as a novel mechanism for hepatocarcinogenesis and hepatic fibrosis/cirrhosis. Therefore, we hypothesize that the hedgehog inhibitor may be an ideal drug target for treating both hepatocellular carcinoma (HCC) and Child-Pugh A cirrhosis (CPA).

DETAILED DESCRIPTION:
This is an open-label, single institution, Phase I, 3+3 dose escalation study of LDE225 in patients with advanced or metastatic hepatocellular carcinoma and Child-Pugh A Cirrhosis who are intolerant to sorafenib. The investigational treatment cycle (21 days) will consist of daily oral LDE225.

Dose escalation will be performed in serial patient cohorts. Up to six patients can be studied at each dose level. Safety and clinical data will be tabulated and the decision to open the next cohort level will be the responsibility of the principal investigator. Dose escalation will be based on the dose-limiting toxicities encountered through Day 42 of investigational treatment.

Patients will be dosed on a flat scale of daily dosing of LDE225 prescribed by the dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pathological confirmation of advanced or metastatic HCC
* HCC not amenable to surgical resection, liver transplantation, chemoembolization, or ablation therapy
* Patients with Child-Pugh A and Child-Pugh B7 (if due to low albumin but not elevated INR or bilirubin) cirrhosis are allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* At least one measurable site of disease (as defined by Response Evaluation Criteria in Solid Tumors)
* Patients with adequate bone marrow, liver and renal function
* Inability to tolerate first-line treatment with sorafenib
* Patient amenable to liver tumor biopsy

Exclusion Criteria:

* Child-Pugh B or Child-Pugh C cirrhosis
* Patients with known Gilbert's Syndrome
* Ongoing alcohol use or abuse defined as > an average of 2 alcoholic beverages daily
* Patients who have had major surgery within 4 weeks of initiation of study medication
* Patients with known brain metastases
* Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study
* Patients with known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* Patients with Hepatitis B and/or Hepatitis C infection are excluded if they are on any of the following viral suppressive agents: boceprevir (Victrelis), ribavirin (Rebetol, Ribatab, Ribasphere), telaprevir (Incivek)
* Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes
* Patients who have previously been treated with systemic LDE225 or with other Hh pathway inhibitors
* Patients who have neuromuscular disorders or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis
* Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment
* Patients who have taken part in an experimental drug study within 4 weeks of initiating study treatment with LDE225
* Patients who are receiving other anti-neoplastic therapy concurrently or within 2 weeks of starting study treatment with LDE225
* Patients who are receiving any anti-coagulation or anti-platelet therapy
* Patients who are receiving treatment with medications known to be strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4/5) or drugs metabolized by cytochrome P450 2B6 (CYP2B6) or cytochrome P450 2C9 (CYP2C9) that have narrow therapeutic index, and that cannot be discontinued before starting study treatment with LDE225
* Impaired cardiac function or clinically significant heart disease
* Patients with contraindications for MRI and/or MRI contrast agents
* Pregnant or nursing (lactating) women
* Women of child-bearing potential must use highly effective contraception during the study and through 6 months after the final dose of study treatment
* Sexually active males who are unwilling to use a condom during intercourse while taking drug and for 6 months after stopping investigational medications and agree not to father a child in this period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities | occurring within 42 days of investigational treatment
  A dose limiting toxicity is a clinically significant adverse event (AE) occurring within 42 days of investigational treatment that is considered by the investigator to be possibly, probably, or definitely related to LDE225.

CONTACTS AND LOCATIONS:
Overall Officials: Jason K. Sicklick, MD, Principal Investigator — University of California Medical Center
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States